CLINICAL TRIAL: NCT01961492
Title: Single Fecal Microbiota Transplantation Via Colonoscope as an Adjunct Therapy in the Treatment of Ulcerative Colitis
Brief Title: Fecal Microbiota Transplantation in Patients With Ulcerative Colitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems in recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Marko Kalliomäki, Specialist, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15881
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fecal microbiota transplantation (Active Comparator): A single fecal microbiota transplantation via colonoscope as an adjunct therapy to standard medical treatment
  Interventions: Other: Fecal microbiota transplantation
- Standard medical treatment (No Intervention): Standard medical treatment as recommended by the ECCO Guidelines of UC therapy.

INTERVENTIONS:
Other: Fecal microbiota transplantation — A single fecal microbiota transplantation through colonoscope
  Arms: Fecal microbiota transplantation

SUMMARY:
The purpose of this study is to find out whether a single fecal microbiota transplantation is an effective and safe treatment as an adjunct to standard therapy in patients with ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* active ulcerative colitis (PUCAI 10-64) in whom fecal microbiota transplantation via colonoscope can be performed

Exclusion Criteria:

* severe ulcerative colitis (PUCAI > 65)

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Activity of ulcerative colitis | Within 1 year after the intervention
  Change from baseline in the Pediatric Ulcerative Colitis Activity Index (PUCAI) at 1 month, 3 months, 6 months, and 12 months.

SECONDARY OUTCOMES:
Colonic inflammation | Within 1 year after the intervention
  Change from baseline in the fecal calprotectin at 1 month, 3 months, 6 months, and 12 months.
Colonic inflammation | Within 1 year after the intervention
  Endoscopic Mayo score at 3 and 12 months after the intervention
Adverse events | Within 1 year after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marko Kalliomäki, MD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland